CLINICAL TRIAL: NCT02856815
Title: Randomized, Open-label, Multi-center and Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of 'Immuncell-LC Group' and 'Non-treatment Group' in the Patients Undergone TACE for Intermediate Stage Hepatocellular Carcinoma
Brief Title: Safety and Efficacy of "Immuncell-LC" in TACE Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILC-IIT-05
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Immuncell-LC; Transarterial Chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immuncell-LC group (Experimental): Adjuvant adoptive immune therapy using a CIK cell agent(Immuncell-LC) 12 times(5 treatments at a frequency of once per week, followed by 5 treatments every 2 weeks, and finally 2 treatments every 4 weeks.
  Interventions: Biological: Immuncell-LC
- Non-treatment group (No Intervention): Non-treatment

INTERVENTIONS:
Biological: Immuncell-LC — Activated T lymphocyte : intravenous dripping of 200ml (1 x 10^9 ~ 2 x 10^10 lymphocytes / 60kg adult) for 1 hour
  Arms: Immuncell-LC group

SUMMARY:
To evaluate the efficacy and safety of 'Immuncell-LC group' and 'non-treatment group' in the patients undergone Transarterial Chemoembolization for intermediate stage hepatocellular carcinoma

DETAILED DESCRIPTION:
ILC-IIT-05 is randomized, open-label, multi-center phase 2 clinical trial. To confirm clinical efficacy and safety between 'Immuncell-LC group' and 'non-treatment group', primary outcome, recurrence free survival(RFS) will be evaluated.

For secondary outcome, overall survival(OS), changes of Alpha Feto Protein(AFP), correlation of between myeloid-derived suppressor cell change and prognosis, adverse event, ECOG-PS and hematological examination will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have consented to the study by providing signature of self
* Patients who are more than 20 and less than 80 years old
* Child-Pugh Class should be A(score 5-6) or B(score 7-8)
* ECOG Performance Status (ECOG-PS) score is less than 1 or equal to
* Patients who have been diagnosed with BCLC stage B hepatocellular carcinoma by pathological/radiological test(Dynamic contrast-enhanced CT or Dynamic MRI) and tumor removal has been confirmed after TACE (When patients have been diagnosed with recurrence of hepatocellular carcinoma after surgery or local treatment, if conditions are same as above, patients could be included)
* Patients who satisfy the following conditions of the blood test and kidney, liver function test

  * Absolute neutrophil count > 500/µL
  * Hemoglobin ≥ 8.5 g/dL
  * Platelet count > 50,000/µL
  * Blood Creatinine ≤ 1.5xupper normal limit
  * Total bilirubin < 3mg/dL
  * Albumin ≥ 2.8g/dL

Exclusion Criteria:

* Patients who have been confirmed with residual tumor or extrahepatic metastases
* Patients who have lymph node metastases or portal vein, hepatic vein invasion
* Patients who have a history of treatments or are in conditions as below

  * Liver transplantation
  * From Informed consent form sign date, systemic chemotherapy in 4 weeks or ongoing adverse drug reactions from anticancer drug in 6 weeks
  * External beam radiation, immunotherapy, molecular target therapy
  * More than 2 times of systemic chemotherapy
  * Biliary reconstruction or endoscopic biliary treatment
* Patients who have a history of auto-immune diseases (Ex. Rheumatoid Arthritis, Systemic Lupus Erythematosus, Vasculitis, Multiple sclerosis, Adolescent Insulin-Dependent Diabetes Mellitus, etc.)
* Patients who have a history of malignant tumors in the recent 5 years prior to the study except hepatocellular carcinoma
* Patients who participated in another clinical trial and conducted treatment in 4 weeks or have a plan for administration of another clinical trial treatment since Informed consent form sign date
* Patients who have uncontrollable or serious disease
* Pregnant women or nursing mother
* Patients who intend to get pregnant during the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2020-08-11 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Recurrence Free Survival (RFS) | baseline until 44 weeks, and then every 3 months until the data cut-off date or 12 months from baseline of last subject
  Every 12 weeks from the baseline until 44 weeks, and then every 3 months until the data cut-off date or 12 months from baseline of last subject

SECONDARY OUTCOMES:
Overall Survival (OS) | baseline until 44 weeks, and then every 3 months until the data cut-off date or 12 months from baseline of last subject
  Every 12 weeks from the baseline until 44 weeks, and then every 3 months until the data cut-off date or 12 months from baseline of last subject
Change of Alpha Feto Protein (AFP) level | Every 12 weeks from the baseline until 44 weeks, and then every 3 months until the data cut-off date or 12 months from baseline of last subject
  Every 12 weeks from the baseline until 44 weeks, and then every 3 months until the data cut-off date or 12 months from baseline of last subject
Correlation of between Myeloid-derived Suppressor Cell change and Prognosis | Every 12 weeks from the baseline until 4 weeks after the last dose of immunotherapy
  Every 12 weeks from the baseline until 4 weeks after the last dose of immunotherapy
Adverse event | From the time the patient provided written informed consent until drop-out or the end of the study or at least 4 weeks after the last dose of immunotherapy
  From the time the patient provided written informed consent until drop-out or the end of the study or at least 4 weeks after the last dose of immunotherapy
Eastern Cooperative Oncology Group Performance Status (ECOG-PS) | From the time the patient provided written informed consent until drop-out or the end of the study or 4 weeks after the last dose of immunotherapy
  From the time the patient provided written informed consent until drop-out or the end of the study or 4 weeks after the last dose of immunotherapy
Hematological examination | Every 12 weeks from the baseline until 4 weeks after the last dose of immunotherapy
  Every 12 weeks from the baseline until 4 weeks after the last dose of immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hwan Yoon, MD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul St.Mary's Hospital, Seoul, Banpo-daero 222 / Seocho-go
  - Seoul National University Hospital, Seoul, Daehak-ro 101/Jongno-gu
  - Severance Hospital, Seoul, Seoul,50-1 Yonsei-ro/Seodaemun-gu

IPD SHARING:
Plan to Share IPD: No